CLINICAL TRIAL: NCT07202988
Title: Investigating the Role of Potatoes in Boosting Vegetable Enjoyment and Consumption Among Adolescents and Emerging Adults
Brief Title: Tasting Plant Forward Meals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Maksi (Other)
Collaborators: Alliance for Potato Research and Education (Other); Penn State University (Other)
Responsible Party: Sponsor-Investigator, Sara Maksi, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 104540
Record Dates: First submitted 2025-09-08; First posted 2025-10-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-10

CONDITIONS: Dietary Exposure
Keywords: Diet Quality; Vegetable Intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potato form 1 (Experimental): The potato served within the vegetable dish will be oil fried.
  Interventions: Other: vegetable combination 1; Other: vegetable combination 2; Other: vegetable combination 3; Other: vegetable combination 4; Other: vegetable combination 5
- Potato form 2 (Experimental): The form of the potato within the vegetable dish will be air fired.
  Interventions: Other: vegetable combination 1; Other: vegetable combination 2; Other: vegetable combination 3; Other: vegetable combination 4; Other: vegetable combination 5

INTERVENTIONS:
Other: vegetable combination 1 — consume 5 consecutive lunch meals, separated by at least one week, that differ in the presence and amount of potato and non-starchy vegetable
Other: vegetable combination 2 — consume 5 consecutive lunch meals, separated by at least one week, that differ in the presence and amount of potato and non-starchy vegetable
Other: vegetable combination 3 — consume 5 consecutive lunch meals, separated by at least one week, that differ in the presence and amount of potato and non-starchy vegetable
Other: vegetable combination 4 — consume 5 consecutive lunch meals, separated by at least one week, that differ in the presence and amount of potato and non-starchy vegetable
Other: vegetable combination 5 — consume 5 consecutive lunch meals, separated by at least one week, that differ in the presence and amount of potato and non-starchy vegetable

SUMMARY:
This study aims to examine how the amount of potato and form of potato within a meal impacts intake and acceptability of other non-starchy vegetables.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-25 years

Exclusion Criteria:

* unable to complete all study procedures
* food allergies to any of the study food

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in liking of non-starchy vegetables served within the plant forward meal | Baseline and after each meal condition (approximately 5 weeks)
  Ranking of degree of liking for each vegetable served within the plat forward meal on a scale of 1-100 on a visual analog scale where 1= extremely dislike to 100= Extremely like. Measured at baseline, within a taste test before each meal, and after each meal.
Differences in total non-starchy vegetable intake between meal conditions | Baseline and after each meal condition (approximately 5 weeks)
  Gram intake of non-starchy vegetable intake at each meal

SECONDARY OUTCOMES:
Adolescent and young adult (18-25 years) knowledge and attitudes of potato nutrition and preparation | After final 5th meal (approximately 5 weeks)
  A series of 10 questions related to nutrient content and health attitude statements where participants rate their agreement on a 1-100 point visual analog scale where 1 = extremely disagree and 100 is extremely agree. Scores will be reported as two subscales -1) knowledge and 2) attitudes with higher scores equating to greater knowledge and more positive attitudes respectively.

OTHER OUTCOMES:
Differences in post meal satiety within person between meal conditions and group differences | After each meal (approximately 5 weeks)
  using ecological momentary assessment to measure hunger, fullness and desire to consume foods on a 1-100 point visual analog scale with 1= not at all to 100=very much

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No